CLINICAL TRIAL: NCT02331160
Title: Rebozo Som Vendingsmetode Ved sædepræsentation (in Danish)
Brief Title: Rebozo and External Cephalic Version in Breech Presentation.
Acronym: RECeiVe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jacob Alexander Lykke, Ass. professor, consultant, MD PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-4-2014-101
Record Dates: First submitted 2014-12-21; First posted 2015-01-06 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Breech Presentation
Keywords: Pregnancy; Breech Presentation; Version, fetal; Musculoskeletal Manipulations; Medicine, Traditional
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rebozo (Experimental): Intervention by Rebozo
  Interventions: Behavioral: Rebozo
- Control (No Intervention): Standard

INTERVENTIONS:
Behavioral: Rebozo — Shaking of the maternal pelvis by the midwife to increase the spontaneous cephalic version rate in breech presentation.
  Arms: Rebozo

SUMMARY:
Breech presentation occurs in approximately 3-5% of all pregnancies, and breech birth is more complicated and risky for the fetus than births of fetuses in the cephalic position.

Therefore, it is desirable to turn the fetus from breech presentation to cephalic position before labour. This is traditionally done by external cephalic version, where the doctor manually tries to turn the fetus; the success rate of this is approximately 50%, and complications occur in about 0.5%. In addition there is discomfort and pain to the pregnant woman.

The investigators will assess the effect of using the rebozo prior to the external version. Use of rebozo is a recognized technique from Mexico, where the midwife with a scarf 'shake' the pregnant woman's pelvis over several sessions, so the fetus spontaneously turns to cephalic presentation or the external version is facilitated.

There are no known complications associated with the rebozo method. Use of rebozo in breech presentation has never before been studied scientifically, but is used in many places in the world. The investigators are planning an open-labeled randomized controlled study in pregnancies with verified breech or transverse presentation: by lot either standard external cephalic version or preceding rebozo-treatment with subsequent external cephalic version.

The investigators want to assess whether the use of rebozo - either as pre-treatment for external cephalic version or as a catalyst of spontaneous version - will increase the incidence of the cephalic presentations at labour and thus reduce the number of planned caesarean section.

The population will be pregnant women with ultrasound verified breech or transverse presentation;all women who fulfill the local guideline criteria for external cephalic version, can be included. Exclusion criteria are non-Danish speaking or reading.

The recruitment will be conducted by midwife at week 35 in the antenatal care. The study design will be open-labeled randomized controlled. Randomisation is done by "closed envelope method" and stratified by parity. Intervention is rebozo exercises performed over 3-5 days from randomization. In case of persistent breech presentation, the woman is offered standard external cephalic version. The control group will also be offered external cephalic version after 3-5 days from randomization.

The investigators will use source data from existing local databases, "Obstetrics Database" and "version Database", for collecting birth outcome. In all stages of intervention documented electronically by project midwives.

The primary objective is the number of successful versions in total, i.e., after intervention and external cephalic version. We expect to increase the success rate from 50% to 65%, thus requiring 378 women in the study.

Secondary objectives are the number of successful vaginal births with birth in head position and total number of caesarean.

ELIGIBILITY:
Inclusion Criteria:

* Understands Danish in writing.
* Intention of accepting vaginal delivery if cephalic presentation.
* Can be offered standard treatment of external cephalic version according to local guidelines, e.g.:

  * Singleton pregnancy
  * Fetus in breech or transverse position
* The gestational age at randomization must be between 35w+0/7d and 37w+4/7d so that the ECV is no later than 38w+0/7d for parous and 37w + 0/7d for nulliparous women.

Exclusion Criteria:

* Women that cannot be offered external cephalic version according local guideline, e.g.:

  * placenta praevia and vasa praevia.
  * Suspicion of severe fetal growth restriction.
  * Severe preeclampsia.
  * Uterus anomalies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Cephalic presentation | After external cephalic version

SECONDARY OUTCOMES:
Version rate by the intervention only | Before external cephalic version
Version rate by the standard external cephalic version | At the external cephalic version
Rate of cesarean section by intervention and presentation. | In labour
Dystocia in labor in cephalic presentation after version | In labour
  Use of Pitocin, vacuum extraction and time frame.
Inducement of labour | Before labour
Time frames for rupture of membranes, labour, first and second stage labour | In Labour
Number of women having epidural | In labour
Fetal presentation, cephalic rotation and asynclitism | In labour
Vaginal and perineal ruptures after vaginal delivery | Hours after delivery
Neonatal outcome | Up to 28 days after delivery
Woman's experience of intervention and external cephalic version | After intervention, before labour or cesarean section.
Obstetrician's rating of difficulty in performing the external cephalic version | After intervention, before labour or cesarean section.
Major complications | During the study
  Fetal demise, placental abruption, fetal distres (by CTG).

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Alexander Lykke, MD PhD, Principal Investigator — Ass. prof., consultant
Locations (1):
- Hvidovre Hospital, dept. of Obstetrics, Copenhagen, Hvidovre, Denmark